CLINICAL TRIAL: NCT06551935
Title: The Effect of Sleep Hygiene and Sleep Extension on Performance in Soccer Players: a Randomized Controlled Trial
Brief Title: Effect of Sleep Hygiene and Sleep Extension on Performance in Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maia (Other)
Responsible Party: Principal Investigator, Lúcio Cunha, Principal Investigator, University of Maia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UI/BD/151482/2021
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Sleep Extension; Sleep Hygiene; Athletic Performance
MeSH Terms: conditions — Sleep Hygiene | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Without sleep intervention
  Interventions: Behavioral: Habitual sleep habits without intervention
- Experimental Group (Experimental): Sleep hygiene and sleep extension
  Interventions: Behavioral: Sleep extension and sleep hygiene

INTERVENTIONS:
Behavioral: Habitual sleep habits without intervention — Sleep habits maintenance
  Arms: Control Group
Behavioral: Sleep extension and sleep hygiene — Players will extend their time in bed by 25%, based on their baseline sleep, and adopt sleep hygiene behaviors: relatively fixed sleep schedule; do not lie in bed awake for long periods of time; no caffeine and no alcohol prior to bedtime; avoid heavy meals close to bedtime; sleep environment cool, dark and quiet; low exposure to screen lights before bedtime, only with nightshift mode and low luminosity (avoid high cognitive demanded activities, like gaming); low luminosity near to bedtime; ensure adequate exposure to light in the morning.
  Arms: Experimental Group

SUMMARY:
Sleep is essential for recovery and performance in athletes, yet they often struggle with inadequate sleep duration and quality. Theoretically, strategies such as sleep extension and sleep hygiene could improve sleep and subsequent recovery in athletes, but their effectiveness remains largely unstudied in the literature. This study aimed to analyze the effects of sleep extension and sleep hygiene on physical and cognitive performance in soccer players.

DETAILED DESCRIPTION:
Twenty soccer players will be randomized (1:1 ratio) into intervention and control groups. The study will last 4 weeks, divided into two periods: baseline (2 weeks) and intervention (2 weeks). In the baseline period, the players will maintain their normal routine and their sleep habits will be monitored by actigraphy and sleep diaries. The players physical performance will be assessed by the 30-15 intermittent fitness test, countermovement jump, isometric mid-thigh pull and 30-meter sprint, while the cognitive performance will be assessed with the 3-minute psychomotor vigilance test. During the intervention period, the intervention group will extend their usual time in bed by 25% than their baseline period, and adopt sleep hygiene behaviors, while the control group will maintain their usual sleep routine. The physical performance of the players of both groups will be assessed with the same physical tests of the baseline period at the end of week 1 and week 2.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years old
* Sex: Male
* Football players competed in an official competition, organized by the Portuguese Football - Federation (FPF) or regional football associations

Exclusion Criteria:

* Players who take sleep medication
* Injured players
* Players with clinical sleep problems

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Sleep | 4 weeks
  Night-time sleep will be monitored each night during the data collection period using wrist-worn actigraphy devices (Actigraph LLC wGT3X-BT, Pensacola, USA). Data will be analyzed using company software (ActiLife LLC Pro software v6.13.3, Pensacola, USA). The sampling frequency will be set to 50 Hz, and the epoch of activity counts 60 s. All sleep variables will be determined using the Sadeh's algorithm
30-15 Intermittent Fitness Test | At the end of the baseline period (2 weeks), after one week of sleep extension and sleep hygiene (intervention period) and after two weeks of sleep extension and sleep hygiene (intervention period)
  The 30-15 IFT consists of 30-second shuttle runs interspersed with 15-second periods of passive recovery. The initial running speed is set at 8 km/h for the first 30-second run and increased by 0.5 km/h for each subsequent stage. Participants ran back and forth between 2 lines 40 m apart at a pace dictated by a pre-recorded beep. During the 15-s recovery period, each player walked forward to the nearest of the 3 lines (in the middle or at one end of the running area, depending on where the previous leg was completed) in preparation for the next leg. Players were instructed to complete as many legs as possible, and the test ended when a player could no longer maintain the prescribed running speed or was unable to reach a 3-m zone around each line at the time of the audio signal on 3 consecutive occasions. If a player was unable to complete the stage, their score was recorded as the last stage they successfully completed, and their running speed was recorded as their VIFT.

SECONDARY OUTCOMES:
30-meters sprint test | At the end of the baseline period (2 weeks), after one week of sleep extension and sleep hygiene (intervention period) and after two weeks of sleep extension and sleep hygiene (intervention period)
  The sprint time (seconds) for 15 and 30 m will be recorded using a photocell system (WITTY, Microgate, Bolzano, Italy). Three photocells will be used to assess 15 and 30 m so that both times could be recorded in a single attempt. Subjects will be asked to assume a stationary starting position with the front foot placed 50 cm behind the first cell. Two maximal attempts will be allowed for all tests, with the best result recorded for analysis.
Countermovement jump (CMJ) | At the end of the baseline period (2 weeks), after one week of sleep extension and sleep hygiene (intervention period) and after two weeks of sleep extension and sleep hygiene (intervention period)
  The CMJ will be recorded with optical detection system (Optogait, Microgate, Bolzano, Italy) and performed with the hands placed on the hips, maintaining the extension of the hip, knee and ankle joints during airtime. Depth during countermovement will be standardized for all players and the average height of three attempts will be recorded.
Isometric Mid-thigh pull (IMTP) | At the end of the baseline period (2 weeks), after one week of sleep extension and sleep hygiene (intervention period) and after two weeks of sleep extension and sleep hygiene (intervention period)
  The IMTP will be performed using a force platform (ForceDecks, VALD, Brisbane, Australia). Athletes will adopt a standard power-pulling stance, with the bar height set to half the thigh length (50% of the distance between the greater trochanter and lateral epicondyle of the knee). Knee and hip angles will be set to 130-140°. Athletes will perform the IMTP two times at maximal effort. Athletes will be instructed to pull upward on the bar "as quickly and explosively as possible," maintaining maximal effort for two to three seconds.
3-min Psychomotor Vigilance Test (PVT) | At the end of the baseline period (2 weeks), after one week of sleep extension and sleep hygiene (intervention period) and after two weeks of sleep extension and sleep hygiene (intervention period)
  The PVT is a standard task used to measure reaction time and has been shown to be sensitive to sleep restriction. The PVT is a 3-minute, iPad-based task (Joggle Research software) requiring athletes to concentrate on a red rectangular box on the screen and tap the screen when a yellow timer appeared in the center of the box. The timer stopped once the participant had responded, indicating the response time in milliseconds. The interstimulus interval varied randomly from 1 to 4 seconds. Responses ≤100ms were labeled "false starts" and responses ≥355 ms were labeled "lapses."

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maia, Maia, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: Undecided